CLINICAL TRIAL: NCT07067970
Title: Comparison of the Efficacy and Safety of Dapoxetine, Kegel Exercises, and Acupuncture in the Treatment of Premature Ejaculation: A Randomized, Double-Blind, Placebo-Controlled Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Ali Ihsan Memmi, MD, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2222486777
Record Dates: First submitted 2025-07-06; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Premature Ejaculation
Keywords: premature ejaculation; acupuncture; dapoksetin; kegel; sham-acupuncture
MeSH Terms: conditions — Premature Ejaculation | interventions — Selective Serotonin Reuptake Inhibitors; Acupuncture Therapy; salicylhydroxamic acid; Exercise

STUDY DESIGN:
Intervention Model Description: A Randomized, Double-Blind, Placebo-Controlled Trial
  Participants will be assigned to one of the following five groups for a 12-week intervention period:Dapoxetine Group:Dosage: 30 mg dapoxetine, taken orally 1-3 hours before anticipated sexual activity, with a maximum of 3 doses per week.
  Administration: Provided in blister packs to ensure compliance. Reference: McMahon et al., 2011.
  Placebo Group:Dosage: Placebo tablets identical in appearance and taste to dapoxetine, administered on the same schedule (1-3 hours before sexual activity, maximum 3 doses per week).
  Administration: Provided in identical blister packs.
  Kegel Exercises Group:Protocol: Participants will perform pelvic floor muscle exercises consisting of three sets of 10-15 contractions daily, each held for 5-10 seconds followed by relaxation.
  Training: Participants will receive initial training from a licensed physiotherapist, with weekly follow-up sessions to ensure proper technique and adherence.
Who Masked: Participant, Investigator
Masking Description: Double-blinding will be maintained by ensuring that participants and outcome assessors are unaware of group assignments. Dapoxetine and placebo tablets will be identical in appearance and packaging. Acupuncture and sham acupuncture procedures will use standardized needles to maintain blinding, with sham acupuncture involving superficial needle insertion at non-active points.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Dapoxetine Group: (Experimental): Dosage: 30 mg dapoxetine taken 1-3 hours before sexual activity (maximum 3 doses per week).
  Duration: 12 weeks.
  Interventions: Drug: serotonin reuptake inhibitor (SSRI)
- Placebo Group (Placebo Comparator): Dosage: Placebo tablet identical in appearance and taste to dapoxetine, following the same dosing protocol.
  Duration: 12 weeks.
  Interventions: Drug: Placebo
- Kegel Exercises Group (Experimental): Protocol: Three sets of 10-15 pelvic floor muscle contractions daily, supervised by a physiotherapist.
  Duration: 12 weeks.
  Interventions: Behavioral: Exercise
- Acupuncture Group (Active Comparator): Protocol: Two 30-minute sessions per week using standardized acupuncture points (e.g., CV4, SP6, ST36) by licensed acupuncturists.
  Duration: 12 weeks
  Interventions: Other: Acupuncture
- Sham Acupuncture Group (Sham Comparator): Protocol: Superficial needle application avoiding active acupuncture points, following the same frequency and duration.
  Duration: 12 weeks.
  Interventions: Other: Sham

INTERVENTIONS:
Drug: serotonin reuptake inhibitor (SSRI) — Dapoxetine Group
  Dosage: 30 mg dapoxetine, taken orally 1-3 hours before anticipated sexual activity, with a maximum of 3 doses per week.
  Administration: Provided in blister packs to ensure compliance. Reference: McMahon et al., 2011.
  Arms: Dapoxetine Group:
Drug: Placebo — Dosage: Placebo tablets identical in appearance and taste to dapoxetine, administered on the same schedule (1-3 hours before sexual activity, maximum 3 doses per week).
  Administration: Provided in identical blister packs.
  Arms: Placebo Group
Other: Acupuncture — Protocol: Two 30-minute acupuncture sessions per week, targeting standardized points (e.g., CV4, SP6, ST36) known to influence sexual function and autonomic nervous system regulation.
  Administration: Performed by licensed acupuncturists following a standardized protocol.
  Reference: Sunay et al., 2011.
  Arms: Acupuncture Group
Other: Sham — Sham Acupuncture Group:Protocol: Two 30-minute sessions per week using superficial needle insertion at non-active points to minimize therapeutic effects while maintaining the placebo effect.
  Administration: Performed by licensed acupuncturists to ensure consistency with the active acupuncture group
  Arms: Sham Acupuncture Group
Behavioral: Exercise — Kegel Exercises Group:Protocol: Participants will perform pelvic floor muscle exercises consisting of three sets of 10-15 contractions daily, each held for 5-10 seconds followed by relaxation.
  Training: Participants will receive initial training from a licensed physiotherapist, with weekly follow-up sessions to ensure proper technique and adherence.
  Reference: Pastore et al., 2014.
  Arms: Kegel Exercises Group

SUMMARY:
This study aims to compare the efficacy and safety of dapoxetine, Kegel exercises, acupuncture, and their placebo controls in the treatment of premature ejaculation (PE). PE is a common male sexual dysfunction characterized by ejaculation occurring within one minute of vaginal penetration, causing distress or interpersonal difficulties (Althof et al., 2014). A total of 250 male participants will be randomized into five groups (dapoxetine, placebo, Kegel exercises, acupuncture, sham acupuncture) for a 12-week treatment period followed by a 4-week follow-up. The primary outcome is the increase in intravaginal ejaculation latency time (IELT), with secondary outcomes including the Premature Ejaculation Diagnostic Tool (PEDT) score, Sexual Quality of Life-Male (SQoL-M) score, and adverse effects.

DETAILED DESCRIPTION:
Study OverviewPremature ejaculation (PE) is one of the most prevalent male sexual dysfunctions, affecting approximately 20-30% of men worldwide. It is defined by the International Society of Sexual Medicine (ISSM) as ejaculation occurring within one minute of vaginal penetration, accompanied by a lack of control over ejaculation and resultant distress or interpersonal difficulties (Althof et al., 2014). PE significantly impacts quality of life, self-esteem, and relationship satisfaction. Current treatment options include pharmacological interventions (e.g., dapoxetine, a selective serotonin reuptake inhibitor), behavioral therapies (e.g., Kegel exercises targeting pelvic floor muscles), and complementary approaches (e.g., acupuncture). However, there is a lack of comprehensive studies comparing the efficacy and safety of these interventions in a single trial. This study aims to address this gap by evaluating the efficacy and safety of dapoxetine, Kegel exercises, acupuncture, and their respective placebo controls in a randomized, double-blind, placebo-controlled trial.Study ObjectivesThe primary objective is to compare the efficacy of dapoxetine, Kegel exercises, and acupuncture in increasing intravaginal ejaculation latency time (IELT) in men with PE, relative to placebo and sham controls. Secondary objectives include assessing improvements in PE severity, sexual quality of life, and the safety profile of each intervention. The study hypothesizes that:Dapoxetine, Kegel exercises, and acupuncture will significantly increase IELT compared to their respective placebo/sham groups.

Differences in efficacy will be observed among the active treatment groups. All interventions will demonstrate acceptable safety profiles with minimal adverse effects.

Study DesignThis is a multi-center, randomized, double-blind, placebo-controlled, parallel-group clinical trial. A total of 250 male participants will be enrolled and randomly assigned to one of five groups (50 participants per group) in a 1:1:1:1:1 ratio. The study duration is 24 months, including 6 months for preparation and recruitment, 12 months for intervention and data collection, and 6 months for data analysis and dissemination. The intervention phase lasts 12 weeks, followed by a 4-week follow-up period to assess sustained effects.Randomization and Blinding:Randomization will be performed using a computer-generated random number sequence to ensure balanced allocation across groups.

Double-blinding will be maintained by ensuring that participants and outcome assessors are unaware of group assignments. Dapoxetine and placebo tablets will be identical in appearance and packaging. Acupuncture and sham acupuncture procedures will use standardized needles to maintain blinding, with sham acupuncture involving superficial needle insertion at non-active points.

Study PopulationThe study will recruit 250 men aged 18-50 years diagnosed with PE according to ISSM criteria. Participants will be enrolled from university hospitals and private clinics across multiple centers (specific sites to be determined).Inclusion Criteria:Male, aged 18-50 years.

Diagnosed with lifelong or acquired PE per ISSM criteria (IELT < 2 minutes, lack of ejaculatory control, and associated distress or interpersonal difficulties).

In a stable sexual relationship with a partner for at least 6 months. Willing to provide written informed consent and comply with study procedures.

Exclusion Criteria:Presence of erectile dysfunction (diagnosed via International Index of Erectile Function score < 21).

Severe psychiatric disorders (e.g., major depression, bipolar disorder) or neurological conditions (e.g., multiple sclerosis, Parkinson's disease).

Current use of selective serotonin reuptake inhibitors (SSRIs) or other psychotropic medications.

History of alcohol or substance dependence. Known contraindications to dapoxetine (e.g., hepatic impairment) or acupuncture (e.g., bleeding disorders).

Previous pelvic floor surgery or trauma affecting pelvic floor muscles.

Sample Size Justification:

The sample size of 250 participants (50 per group) was calculated based on a power analysis (α=0.05, power=0.80) to detect a clinically meaningful 30% increase in IELT, assuming a standard deviation derived from prior studies (McMahon et al., 2011). This accounts for an estimated 10% dropout rate.InterventionsParticipants will be assigned to one of the following five groups for a 12-week intervention period:Dapoxetine Group:Dosage: 30 mg dapoxetine, taken orally 1-3 hours before anticipated sexual activity, with a maximum of 3 doses per week.

Administration: Provided in blister packs to ensure compliance. Reference: McMahon et al., 2011.

Placebo Group:Dosage: Placebo tablets identical in appearance and taste to dapoxetine, administered on the same schedule (1-3 hours before sexual activity, maximum 3 doses per week).

Administration: Provided in identical blister packs.

Kegel Exercises Group:Protocol: Participants will perform pelvic floor muscle exercises consisting of three sets of 10-15 contractions daily, each held for 5-10 seconds followed by relaxation.

Training: Participants will receive initial training from a licensed physiotherapist, with weekly follow-up sessions to ensure proper technique and adherence.

Reference: Pastore et al., 2014.

Acupuncture Group:Protocol: Two 30-minute acupuncture sessions per week, targeting standardized points (e.g., CV4, SP6, ST36) known to influence sexual function and autonomic nervous system regulation.

Administration: Performed by licensed acupuncturists following a standardized protocol.

Reference: Sunay et al., 2011.

Sham Acupuncture Group:Protocol: Two 30-minute sessions per week using superficial needle insertion at non-active points to minimize therapeutic effects while maintaining the placebo effect.

Administration: Performed by licensed acupuncturists to ensure consistency with the active acupuncture group.

Outcome MeasuresPrimary Outcome Measure:Intravaginal Ejaculation Latency Time (IELT): Measured by stopwatch during sexual intercourse, reported as the weekly average. Participants will record IELT for each sexual encounter. Time points: Baseline, Week 4, Week 8, Week 12, and Follow-up (Week 16).

Secondary Outcome Measures:Premature Ejaculation Diagnostic Tool (PEDT): A validated 5-item questionnaire assessing PE severity, including control, frequency, and distress (Symonds et al., 2007). Time points: Baseline, Week 4, Week 8, Week 12, and Follow-up (Week 16).

Sexual Quality of Life-Male (SQoL-M): A validated scale measuring the impact of sexual dysfunction on quality of life (Abraham et al., 2008). Time points: Baseline, Week 4, Week 8, Week 12, and Follow-up (Week 16).

Adverse Effects: Any adverse events (e.g., nausea, headache, skin irritation) will be systematically recorded using a standardized adverse event reporting form throughout the study.

Data Collection and ManagementIELT Measurement: Participants will use a stopwatch to record IELT during sexual intercourse and report weekly averages via a secure electronic diary.

Questionnaires: PEDT and SQoL-M will be administered electronically or on paper at specified time points.

Adverse Events: Participants will report adverse effects at each study visit, with additional spontaneous reporting encouraged via a dedicated contact line.

Data Management: Data will be stored in a secure, anonymized database compliant with data protection regulations (e.g., GDPR). Regular audits will ensure data integrity.

Statistical AnalysisPrimary Outcome (IELT): Analyzed using repeated-measures ANOVA with post-hoc tests to compare changes in IELT across groups and time points.

Secondary Outcomes (PEDT, SQoL-M): Analyzed using the Kruskal-Wallis test for non-parametric data, with pairwise comparisons as needed.

Adverse Effects: Analyzed using Chi-square tests to compare the frequency and severity of adverse events across groups.

Significance Level: p<0.05. Software: Statistical analysis will be conducted using SPSS (version 28) or R (version 4.3 or higher).

Handling Missing Data: Intention-to-treat analysis will be used, with last observation carried forward (LOCF) for missing data points.

Ethical ConsiderationsThe study will adhere to the principles of the Declaration of Helsinki and Good Clinical Practice (GCP) guidelines.

Approval will be obtained from local Institutional Review Boards (IRBs) at each participating site.

All participants will provide written informed consent after receiving detailed information about the study's purpose, procedures, risks, and benefits.

Participant confidentiality will be ensured through anonymization of data and secure storage.

A Data and Safety Monitoring Board (DSMB) will oversee the study to ensure participant safety and protocol adherence.

Study TimelineMonths 0-2: Obtain IRB approval, finalize study sites, and train personnel.

Months 3-6: Recruit and randomize participants. Months 7-18: Conduct interventions and collect data (12-week intervention + 4-week follow-up).

Months 19-24: Analyze data, prepare manuscripts, and disseminate results.

Expected ResultsThe study anticipates that dapoxetine and acupuncture will significantly increase IELT compared to their placebo/sham controls, with Kegel exercises potentially showing sustained effects during the follow-up period. Improvements in PEDT and SQoL-M scores are expected in active treatment groups, reflecting enhanced ejaculatory control and sexual quality of life. Adverse effects are expected to be minimal, with dapoxetine potentially associated with mild side effects (e.g., nausea, headache) and acupuncture with minor local reactions (e.g., bruising).LimitationsSelf-reported measures (IELT, PEDT) may introduce subjectivity, despite the use of validated tools.

Sham acupuncture may not fully eliminate placebo effects, potentially reducing the observed effect size.

The 16-week follow-up period may limit insights into the long-term efficacy of interventions.

Participant adherence to Kegel exercises may vary, though supervised training aims to mitigate this.

Dissemination PlanResults will be submitted for publication in peer-reviewed journals, such as The Journal of Sexual Medicine or European Urology, and presented at international conferences (e.g., ISSM or EAU meetings). A summary of findings will be shared with participants and made publicly available on clinicaltrials.gov upon study completion.ReferencesAlthof, S. E., et al. (2014). An update of the International Society of Sexual Medicine's guidelines for the diagnosis and treatment of premature ejaculation (PE). The Journal of Sexual Medicine, 11(6), 1392-1422.

McMahon, C. G., et al. (2011). Efficacy and safety of dapoxetine for the treatment of premature ejaculation: Integrated analysis of results from five phase 3 trials. The Journal of Sexual Medicine, 8(2), 524-539.

Pastore, A. L., et al. (2014). Pelvic floor muscle rehabilitation for patients with lifelong premature ejaculation: A novel therapeutic approach. Therapeutic Advances in Urology, 6(3), 83-88.

Sunay, D., et al. (2011). Acupuncture versus paroxetine for the treatment of premature ejaculation: A randomized, placebo-controlled clinical trial. European Urology, 59(5), 765-771.

Symonds, T., et al. (2007). Development and validation of a premature ejaculation diagnostic tool. European Urology, 52(2), 565-573.

Abraham, L., et al. (2008). Development and validation of a quality-of-life measure for men with sexual dysfunction. Quality of Life Research, 17(4), 575-585.

ELIGIBILITY:
Inclusion Criteria:

* Male, aged 18-50 years. Diagnosed with lifelong or acquired PE per ISSM criteria (IELT < 2 minutes, lack of ejaculatory control, and associated distress or interpersonal difficulties).

In a stable sexual relationship with a partner for at least 6 months. Willing to provide written informed consent and comply with study procedures.

Exclusion Criteria:

* Presence of erectile dysfunction (diagnosed via International Index of Erectile Function score < 21).

Severe psychiatric disorders (e.g., major depression, bipolar disorder) or neurological conditions (e.g., multiple sclerosis, Parkinson's disease).

Current use of selective serotonin reuptake inhibitors (SSRIs) or other psychotropic medications.

History of alcohol or substance dependence. Known contraindications to dapoxetine (e.g., hepatic impairment) or acupuncture (e.g., bleeding disorders).

Previous pelvic floor surgery or trauma affecting pelvic floor muscles.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — premature ejaculation is male condition
Enrollment: 250 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Intravaginal Ejaculation Latency Time (IELT): | Time points: Baseline, Week 4, Week 8, Week 12, and Follow-up (Week 16
  Measured by stopwatch during sexual intercourse, reported as the weekly average. Participants will record IELT for each sexual encounter.

SECONDARY OUTCOMES:
Premature Ejaculation Diagnostic Tool (PEDT): | Time points: Baseline, Week 4, Week 8, Week 12, and Follow-up (Week 16).
  A validated 5-item questionnaire assessing PE severity, including control, frequency, and distress (Symonds et al., 2007).

CONTACTS AND LOCATIONS:
Locations (1):
- Medipol, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
not decided yet

REFERENCES:
- [Background] Sunay D, Sunay M, Aydogmus Y, Bagbanci S, Arslan H, Karabulut A, Emir L. Acupuncture versus paroxetine for the treatment of premature ejaculation: a randomized, placebo-controlled clinical trial. Eur Urol. 2011 May;59(5):765-71. doi: 10.1016/j.eururo.2011.01.019. Epub 2011 Jan 18. PMID 21256670
- [Background] Pastore AL, Palleschi G, Fuschi A, Maggioni C, Rago R, Zucchi A, Costantini E, Carbone A. Pelvic floor muscle rehabilitation for patients with lifelong premature ejaculation: a novel therapeutic approach. Ther Adv Urol. 2014 Jun;6(3):83-8. doi: 10.1177/1756287214523329. PMID 24883105
- [Background] McMahon CG, Althof SE, Kaufman JM, Buvat J, Levine SB, Aquilina JW, Tesfaye F, Rothman M, Rivas DA, Porst H. Efficacy and safety of dapoxetine for the treatment of premature ejaculation: integrated analysis of results from five phase 3 trials. J Sex Med. 2011 Feb;8(2):524-39. doi: 10.1111/j.1743-6109.2010.02097.x. Epub 2010 Nov 8. PMID 21059176
- [Background] Althof SE, McMahon CG, Waldinger MD, Serefoglu EC, Shindel AW, Adaikan PG, Becher E, Dean J, Giuliano F, Hellstrom WJ, Giraldi A, Glina S, Incrocci L, Jannini E, McCabe M, Parish S, Rowland D, Segraves RT, Sharlip I, Torres LO. An Update of the International Society of Sexual Medicine's Guidelines for the Diagnosis and Treatment of Premature Ejaculation (PE). Sex Med. 2014 Jun;2(2):60-90. doi: 10.1002/sm2.28. PMID 25356302